CLINICAL TRIAL: NCT05875181
Title: Examining the Impact of Transcranial Focused Ultrasound (tFUS) on Reward Neural Circuitry
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The data from this pilot study was intended to generate effect sizes and pilot data for a subsequent grant application. However, the grant application was awarded funding before this pilot study collected data.
Sponsor: Mary Phillips, MD MD (Cantab) (Other)
Responsible Party: Sponsor-Investigator, Mary Phillips, MD MD (Cantab), Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY23020148
Record Dates: First submitted 2023-04-24; First posted 2023-05-25 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Impulsive Behavior
Keywords: transcranial focused ultrasound; Magnetic Resonance Imaging
MeSH Terms: conditions — Impulsive Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- VS tFUS/Sham tFUS (Experimental): VS tFUS (tFUS applied to the ventral striatum) Sham tFUS (go through the motions of applying tFUS to the VS)
  Interventions: Device: tFUS; Device: Sham tFUS
- Sham tFUS/VS tFUS (Experimental): VS tFUS (tFUS applied to the ventral striatum) Sham tFUS (go through the motions of applying tFUS to the VS)
  Interventions: Device: tFUS; Device: Sham tFUS

INTERVENTIONS:
Device: tFUS — tFUS is a brief stimulation of a part of the brain called the ventral striatum with low-intensity sound waves that pass through the scalp and skull safely.
Device: Sham tFUS — Sham tFUS goes through the motions of applying tFUS to the brain. Participants will know that one session will be a sham, but they will be blinded to which session is the sham

SUMMARY:
The investigators aim to examine the immediate effect of transcranial focused ultrasound (tFUS) on brain activity and emotions in healthy adults as a first stage toward understanding the predisposing brain mechanisms of underlying substance use disorders.

DETAILED DESCRIPTION:
In a small pilot study the investigators propose to demonstrate feasibility of using tFUS to target the ventral striatum (VS) in humans by examining VS target engagement by tFUS in healthy human volunteers using a reward processing task that reliably activates the VS.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years of age
* No psychiatric history

Exclusion Criteria:

* Not between 18-35 years of age
* Has psychiatric history
* History of head injury, neurological, pervasive developmental disorder (e.g. autism), systemic medical disease and treatment (medical records, participant report)
* Mini-Mental State Examination (MMSE) score (cognitive state) <24
* Premorbid North American Adult Reading Test (NAART) intelligent quotient (IQ) estimate<85
* Visual disturbance: <20/40 Snellen visual acuity
* Left/mixed handedness (Annett criteria)
* History of alcohol/substance use disorder (SUD) (all substances, including nicotine), and/or illicit substance use (except cannabis) over the last 6 months (Structured Clinical Interview for Diagnostic and Statistic Manual of Mental Disorders , 5th Edition (DSM-5) (SCID-5)). Urine tests on scan days will exclude current illicit substance use (except cannabis). Salivary alcohol tests on scan days will exclude intoxicated individuals
* Magnetic resonance imaging (MRI) exclusion: metallic objects, e.g., surgical implants; claustrophobia; positive pregnancy test for females or self-report pregnancy
* Unable to understand English
* Individuals with a positive pregnancy test will be excluded from the study and not undergo a computerized tomography (CT) scan or MRI scan
* Present or history of seizure disorder

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06-19 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Blood oxygen level-dependent (BOLD) signal | 30-60 minutes
  The blood oxygen level-dependent (BOLD) signal indicates brain activity and connectivity

CONTACTS AND LOCATIONS:
Overall Officials: Mary Phillips, MD, MD, Principal Investigator — University of Pittsburgh; Fabio Ferrarelli, MD, PhD, Principal Investigator — University of Pittsburgh; Khaled Moussawi, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Informed consent will be collected from study participants that allows for broad sharing of participants' de-identified data. Data transfer procedures will be in accordance with all Institutional Review Board guidelines and federal regulations including HIPAA (Health Insurance Portability and Accountability Act of 1996).
Time Frame: The principal investigators (PIs) reserve the right to publish on the stated aims in a timely manner. Data will be available for addressing other research questions (i.e. which are not described in funded/pending grants) as soon as the data have been checked for accuracy (a period which will be no later than one year after the completion of each assessment). After the study has ended, the study investigators will continue to test the stated aims, but will also continue to solicit collaborations with outside researchers and to consider data requests in a timely manner.
Access Criteria: Outside investigators must submit a 1)proposal of the study aims, hypotheses, variables/constructs, analytic approach, and estimated duration of the proposed research; 2)resume, qualifications, source of financial support, and conflict of interest statement; 3)sign a data-sharing agreement and confidentiality statement that stipulates using the data for the stated research purposes only, securing the data using appropriate computer technology, not manipulating the data in order to identify participants, acknowledging the grant that supported data collection and management in publications/presentations, and destroying or returning the data after analyses are complete; 4)obtain approval from their Institutional Review Board, and along with other staff members who have access to the data, submit certificates of the University of Pittsburgh Education and Certification Program in Research Practice Fundamentals or provide written documentation pf similar human subjects protection training.